CLINICAL TRIAL: NCT00909480
Title: A 26 Week Randomised, Multinational, Open Labelled, 2 Armed, Parallel Group, Treat-to-target Once Daily Treatment Trial With Insulin Detemir Versus Insulin Glargine, Both in Combination With Metformin in Subjects With Type 2 Diabetes
Brief Title: Effect of Insulin Detemir and Insulin Glargine on Blood Glucose Control in Subjects With Type 2 Diabetes
Acronym: EFFICACY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1768
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDet (Experimental): Individually adjusted insulin detemir once daily + metformin at least 1500 mg/day
  Interventions: Drug: insulin detemir
- IGlar (Active Comparator): Individually adjusted insulin glargine once daily + metformin at least 1500 mg/day
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin detemir — Treat-to-target (individually adjusted dose) titration according to titration algorithm.
  S.c. (under the skin) injection once daily as an add-on to subjects' stable pre-trial metformin dose (at least 1500 mg/day). Any other use of OAD will be discontinued
  Arms: IDet
Drug: insulin glargine — Treat-to-target (individually adjusted dose) titration according to titration algorithm.
  S.c. (under the skin) injection once daily as an add-on to subjects' stable pre-trial metformin dose (at least 1500 mg/day). Any other use of OAD will be discontinued
  Arms: IGlar

SUMMARY:
This trial is conducted in Asia, South America and the United States of America (USA).

The aim of this clinical trial is to determine whether two insulin treatments given once daily are equally effective with respect to the blood glucose lowering effect in subjects with type 2 diabetes inadequately controlled on metformin treatment with or without an additional anti-diabetic drug (OAD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for at least 6 months
* Stable treatment with a total daily dose of at least 1500 mg metformin or maximum tolerated dose (minimum 1000 mg) with or without one other OAD (sulphonylureas, meglitinides, thiazolidinediones or dipeptidyl peptidase-4 (DPP-4) inhibitors) for at least 3 months
* Subject is insulin-naive (short-term insulin treatment of up to 14 days is allowed)
* HbA1c (glycosylated haemoglobin) 7.0-9.0 % (both inclusive) by central laboratory analysis (one re-test within one week is allowed)
* Body Mass Index (BMI) less than or equal to 35.0 kg/m^2

Exclusion Criteria:

* Any contraindication to insulin detemir or insulin glargine according to the local labelling
* Receipt of any investigational product within 4 weeks
* Anticipated change of dose of any systemic treatment with products, which in the Investigator's opinion could interfere with glucose metabolism (e.g. systemic corticosteroids)
* Clinically significant diseases which, in the Investigator's opinion may confound the results of the trial or pose additional risk in administering trial product
* Any other condition that the Investigator feels would interfere with trial participation or evaluation of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (77):
- United States (66):
  - Novo Nordisk Investigational Site, Litchfield Park, Arizona
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Escondido, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Redlands, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Spring Valley, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Hollywood, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Ocala, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Winter Haven, Florida
  - Novo Nordisk Investigational Site, Powder Springs, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Independence, Kansas
  - Novo Nordisk Investigational Site, Shawnee Mission, Kansas
  - Novo Nordisk Investigational Site, Portland, Maine
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Clilfton, New Jersey
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Cayahoga Falls, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Gallipolis, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Clarion, Pennsylvania
  - Novo Nordisk Investigational Site, Lancaster, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Taylors, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Martinsburg, West Virginia
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Mar del Plata
- India (3):
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Thriruvananthapuram
- Puerto Rico (2):
  - Novo Nordisk Investigational Site, Manatí
  - Novo Nordisk Investigational Site, Trujillo Alto
- Novo Nordisk Investigational Site, Seoul, South Korea
- Thailand (2):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Pathum Thani

REFERENCES:
- [Result] Meneghini L, Kesavadev J, Demissie M, Nazeri A, Hollander P. Once-daily initiation of basal insulin as add-on to metformin: a 26-week, randomized, treat-to-target trial comparing insulin detemir with insulin glargine in patients with type 2 diabetes. Diabetes Obes Metab. 2013 Aug;15(8):729-36. doi: 10.1111/dom.12083. Epub 2013 Mar 13. PMID 23421331
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were a total of 85 trial sites in 5 countries: 70 in the United States of America (USA), 5 in Thailand, 4 in Korea, 2 in India and 4 in Argentina
Pre-assignment Details: After randomisation, the dose and dosing frequency of metformin were maintained throughout the trial in both treatment arms. Other oral anti-diabetic drug (OAD) was discontinued before use of trial product
Period: Overall Study
Arm/Group | IDet | IGlar
Started | 228 | 229
Exposed | 226 (2 subjects withdrew before exposure to trial insulin) | 227 (2 subjects withdrew before exposure to trial insulin)
Completed | 190 | 188
Not Completed | 38 | 41
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 6 | 8
Not completed — Withdrawal criteria | 9 | 11
Not completed — Unclassified | 18 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDet | IGlar | Total
Number analyzed (Participants) | 226 | 227 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.2) | 57.3 (10.3) | 57.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 101 | 198
  Male | 129 | 126 | 255
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian/Alaska Native | 2 | 0 | 2
  Asian | 56 | 60 | 116
  Black/African American | 22 | 31 | 53
  Native Hawaiian or pacific islander | 1 | 0 | 1
  White | 138 | 129 | 267
  Other | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 51 | 56 | 107
  Not Hispanic or Latino | 164 | 150 | 314
  Not Applicable | 11 | 21 | 32
Weight [Mean (Standard Deviation); unit: kg] | 82.8 (17.2) | 81.7 (16.2) | 82.3 (16.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.86 (3.96) | 29.06 (3.9) | 28.96 (3.93)
HbA1c (Glycosylated haemoglobin A1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 7.96 (0.62) | 7.86 (0.58) | 7.91 (0.6)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.66 (2.26) | 8.46 (2.21) | 8.56 (2.24)
Region of Enrolment [Number; unit: participants]
  Argentina | 11 | 10 | 21
  India | 19 | 32 | 51
  Korea, Republic of | 16 | 10 | 26
  Thailand | 17 | 16 | 33
  United States | 163 | 159 | 322
Height [Mean (Standard Deviation); unit: meters] | 1.69 (0.11) | 1.67 (0.1) | 1.68 (0.11)
Stratification [Number; unit: participants]
  Metformin+thiazolidinedione (TZD) | 15 | 15 | 30
  Metformin + other OAD other than TZD | 149 | 150 | 299
  Metformin monotherapy | 62 | 62 | 124
Diabetes History [Mean (Standard Deviation); unit: years] | 7.99 (5.56) | 8.44 (6.56) | 8.22 (6.08)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline
Time Frame: Week 0, Week 26
Population: Full analysis set: All randomised subjects exposed to at least one dose of trial product categorised by randomised treatment.
Measure: Mean (Standard Deviation); unit: percentage point change
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 203
percentage point change | -0.48 (0.94) | -0.74 (0.76)
Statistical Analysis 1: Comparison: IDet vs IGlar; Test type: Non-Inferiority or Equivalence — Non-inferiority margin: 0.4%; ANCOVA; Full analysis set, Model adjusted for: HbA1c at baseline, previous oral anti-diabetic treatment and country; Mean Difference (Net) = 0.3003, 95% CI [0.1427 to 0.4580]

2. Secondary Outcome: Percentage of Subjects Achieving HbA1c Less Than or Equal to 7.0%
Description: The percentage of subjects - overall and by previous OAD treatment - meeting the HbA1c less than or equal to 7%
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 204
percentage of subjects
  Metformin monotherapy | 55 | 70
  Metformin+TZD | 40 | 40
  Metformin+2nd OAD other than TZD | 31 | 47
  All | 38 | 53

3. Secondary Outcome: Percentage of Subjects Achieving HbA1c of 7% or Less With no Hypoglycaemia
Description: The subjects must have reached target and not have experienced any confirmed symptomatic hypoglycaemia or any confirmed major hypoglycaemia within the last 30 days of treatment.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 204
percentage (%) of subjects
  Metformin monotherapy | 48 | 52
  Metformin+TZD | 33 | 33
  Metformin+2nd OAD other than TZD | 25 | 33
  All | 32 | 38

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Less Than or Equal to 6.5%
Description: The percentage of subjects - overall and by previous OAD treatment - meeting the HbA1c of 6.5% or less
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 204
percentage (%) of subjects
  Metformin monotherapy | 22 | 30
  Metformin+TZD | 13 | 13
  Metformin+2nd OAD other than TZD | 5 | 17
  All | 11 | 21

5. Secondary Outcome: Percentage of Subjects Achieving HbA1c of 6.5% or Less With no Hypoglycaemia
Description: as for outcome 3
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: percentage (%) of subjects
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 204
percentage (%) of subjects
  Metformin monotherapy | 22 | 21
  Metformin+TZD | 7 | 13
  Metformin+2nd OAD other than TZD | 3 | 13
  All | 9 | 15

6. Secondary Outcome: Fasting Plasma Glucose (FPG)
Time Frame: Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 209 | 209
mmol/L | 6.22 (1.88) | 6.09 (2.38)

7. Secondary Outcome: Within-subject Variation of Self Measured Plasma Glucose (SMPG) Before Breakfast
Description: The median values of the sample standard variation (the within subject variation) within the IDet and IGlar arms were plotted against time.
Time Frame: Week 26
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: mmol/L
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
mmol/L
  Metformin Monotherapy | 0.48 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided | 0.67 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided
  Metformin+TZD | 0.72 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided | 0.84 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided
  Metformin+2nd OAD other than TZD | 0.6 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided | 0.71 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided
  Overall | 0.57 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided | 0.71 (NA) — The outcome 'within-subject variation' is defined as the sample standard-deviation of the non-missing pre-breakfast plasma-glucose values on three days before a visit, therefore no additional standard deviation of the standard is provided

8. Secondary Outcome: Glycaemic Control as Measured by Plasma Glucose (9-point Self-measured Profiles)
Description: Plasma glucose measured: before breakfast, 2 hours after breakfast, before lunch, 2 hours after lunch, before dinner, 2 hours after dinner, bedtime and at 3 am.
Time Frame: Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
mmol/L
  Before breakfast (N=200, N=197) | 5.8 (1.5) | 5.9 (1.9)
  2 hours after breakfast (N=192, N=188) | 9.1 (2.9) | 8.7 (2.8)
  Before Lunch (N=193, N=189) | 7.2 (2.8) | 6.6 (2.2)
  2 hours After Lunch (N=194, N=186) | 9.7 (3.2) | 8.8 (2.9)
  Before Dinner (N=194, N=186) | 8.2 (2.6) | 7.5 (2.5)
  2 hours after dinner (N=192, N=190) | 10.3 (3) | 9.8 (2.8)
  Bedtime (N=190, N=183) | 9.5 (3.2) | 9 (3.1)
  At 3AM (N=193, N=186) | 6.6 (2.5) | 6.3 (2.1)
  Before Breakfast Next Day (N=197, N=195) | 5.7 (1.7) | 5.6 (1.7)

9. Secondary Outcome: Incidence of Hypoglycaemic Episodes During the Trial
Description: Number of hypoglycaemic episodes from Week 0 to Week 26, defined as major, minor, or symptoms only. Major if unable to treat her/himself. Minor if able to treat her/himself and plasma glucose below 3.1 mmol/L. Symptoms only if able to treat her/himself and no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: Weeks 0-26
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
episodes
  All Events | 329 | 457
  Major | 0 | 2
  Minor | 119 | 156
  Symptoms only | 210 | 299

10. Secondary Outcome: Hypoglycaemic Episodes, Diurnal
Description: as for outcome 9
Time Frame: Weeks 0-26
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
episodes
  Major | 0 | 2
  Minor | 75 | 118
  Symptoms only | 128 | 222

11. Secondary Outcome: Hypoglycaemic Episodes, Nocturnal
Description: as for outcome 9
Time Frame: Weeks 0-26
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
episodes
  Major | 0 | 0
  Minor | 39 | 30
  Symptoms only | 76 | 61

12. Secondary Outcome: Hypoglycemic Episodes, Unclassifiable
Description: as for outcome 9
Time Frame: Weeks 0-26
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial product.
Measure: Number; unit: episodes
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
episodes
  Major | 0 | 0
  Minor | 5 | 8
  Symptoms only | 6 | 16

13. Secondary Outcome: Change in Body Weight From Baseline
Time Frame: Week 0, Week 26
Population: Safety Analysis Set is all randomised subjects exposed to at least one dose of trial product.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 196 | 193
kg | -0.49 (3.31) | 1 (3.07)

14. Secondary Outcome: Number of Subjects Having the Adverse Event "Incorrect Dose Administered"
Description: Number of subjects having the adverse event "incorrect dose administered" within the system organ class "Injury, poisoning and procedural complications"
Time Frame: Weeks 0-26
Population: Safety Analysis Set: All subjects that received at least one dose of the trial product.
Measure: Number; unit: Subjects
Arm/Group | IDet | IGlar
Number analyzed (Participants) | 226 | 227
Subjects | 12 | 24

ADVERSE EVENTS:
Time Frame: Weeks 0-26
Description: Safety Analysis Set: All subjects that received at least one dose of the trial product.
Arm/Group | IDet | IGlar
Serious Adverse Events (participants affected / at risk) | 7/226 | 12/227
Other Adverse Events (participants affected / at risk) | 26/226 | 18/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDet (N=226) | IGlar (N=227)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Ludwig Angina (Infections and infestations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDet (N=226) | IGlar (N=227)
Nasopharyngitis (Infections and infestations) | 24 (30) | 18 (22)
Upper Respiratory Tract Infection (Infections and infestations) | 18 (19) | 9 (11)
Influenza (Infections and infestations) | 11 (12) | 12 (12)
Diarrhoea (Gastrointestinal disorders) | 16 (19) | 10 (11)
Nausea (Gastrointestinal disorders) | 12 (12) | 5 (5)
Headache (Nervous system disorders) | 17 (40) | 17 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right not to release data before passing specified milestones. This includes the right not to release interim results that may later be found to be incorrect. At the end of the trial, one or more manuscripts will be prepared in collaboration between Investigator(s) and Novo Nordisk. Novo Nordisk will not suppress or veto publications but will reserve the right to postpone publication and/or communication for a short time to protect intellectual property.